CLINICAL TRIAL: NCT04488874
Title: Clinical Effectiveness of Hypertonic Sodium Lactate Infusion for Intraoperative Brain Relaxation in Patients Undergoing Scheduled Craniotomy for Supratentorial Brain Tumor Resection: Study Protocol of a Single Center Double-blind Randomized Controlled Phase II Pilot Trial
Brief Title: Sodium Lactate and Brain Relaxation (LSD)
Acronym: LSD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: API/2017/81
Record Dates: First submitted 2019-04-08; First posted 2020-07-28 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Sodium Lactate; Intracranial Hypertension; Brain Relaxation
Keywords: Brain relaxation; Sodium lactate; Mannitol 20%; Neurosurgery
MeSH Terms: conditions — Intracranial Hypertension | interventions — Sodium Lactate; Mannitol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not known which of Sodium lactate or Mannitol will they receive. The drug will be hidden by an opaque drape during its administration and as soon as the administration is over it will be taken out of the operating room, so the neurosurgeon won't know which drug was given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Lactate (Experimental): Intravenous Molar Sodium Lactate is administered during the first surgical incision. The dose is 2.5mL/kg.
  Interventions: Drug: Sodium Lactate
- Mannitol 20% (Active Comparator): Intravenous mannitol 20% is administered during the first surgical incision. The dose is 5mL/kg (1g/kg).
  Interventions: Drug: Mannitol 20% Infusion

INTERVENTIONS:
Drug: Sodium Lactate — Sodium lactate is administered at 2.5mL/kg during the first surgical incision. Neurosurgeon will evaluate the brain relaxation using a validated scale once the dura is open. A stage 1(perfectly relaxed) or 2((acceptably relaxed) is considered satisfactory.
  Sodium Lactate and Mannitol 20% are used at an equimolar dose
  Arms: Sodium Lactate
Drug: Mannitol 20% Infusion — Mannitol 20% is administered intravenously at a dose of 5mL/kg, so 1g/kg, during the first surgical incision. Neurosurgeon will evaluate the brain relaxation using a validated scale once the dura is open. A stage 1(perfectly relaxed) or 2((acceptably relaxed) is considered satisfactory.
  Arms: Mannitol 20%

SUMMARY:
Resection surgery of brain tumors by craniotomy requires efficient brain relaxation intraoperatively in order to avoid injuries caused by the brain retractors (such as ischemic-reperfusion and cerebral oedema). The gold standard for the brain relaxation during a surgery is Mannitol 20%.

Molar sodium lactate is now used to induce brain relaxation in patients with traumatic brain injury and intracranial hypertension due to its osmotic effect. Furthermore, the injection of sodium lactate may lead to better neuronal metabolism during cerebral aggression, and may participate to the reduction of cerebral oedema and secondary injuries.

LSD is a pilot randomised trial which tries to assess the interest of intravenous administration of molar Sodium Lactate on the quality of brain relaxation in surgical resection of supratentorial brain tumors by craniotomy.

The primary outcome measure is the quality of brain relaxation, evaluated by neurosurgeon at the opening of the dura, by a validated brain relaxation scale.

DETAILED DESCRIPTION:
It's a prospective, comparative, randomised, double blinded study. It will enroll 50 patients undergoing resection surgery of supratentorial brain tumor. They will be randomly divided in 2 groups of 25 patients each : Mannitol 20% and molar Sodium Lactate. The only difference between the 2 groups is the drug used for brain relaxation at the surgical incision : Mannitol or Sodium lactate.

The outcome measures include quality of brain relaxation, need of "rescue" therapy to get an adequate brain relaxation, electrolytes alterations, change in lactate serum level, quantification of post operative brain swelling by MRI, time of extubation, Glasgow Coma Scale, neuropsychological evaluation, blood levels of Protein S100-β, NSE (Neuron-Specific Enolase) and GFAP Glial Fibrillary Acid Protein), morbidity and mortality during 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA 1, ASA 2 ou ASA 3, meaning they don't have any unstable comorbidities which could be a threat to life.
* Scheduled surgery for resection of supratentorial brain tumors by craniotomy under general anesthesia
* Unilateral brain tumor
* Deviation of the falx cerebri > 3mm on the preoperative imaging
* Pharmacological brain relaxation required by the neurosurgeon in charge of the patient.
* Patient who has been informed and who signed the free informed consent to participate to the study. Meaning the patient understood the purpose and the procedures required by the study and agreed to participate and obey the requirements and restrictions of this study.
* Affiliation to a social security system or recipient of a such system.

Exclusion Criteria:

* Emergency surgery
* Age < 18 years old or > 75 years old
* ASA score IV-V
* Legal incapability or limited legal capacity
* Patient who will unlikely cooperate to the study and/or poor cooperation foreseen by the investigator
* Preoperative Glasgow score < 13
* Pregnant woman and/or breastfeeding
* Body index masse< 18 kg.m-2 ou > 30 kg.m-2
* Preoperative hyponatremia < 130mmol/l or hypernatremia > 145 mmol/l
* Osmotherapy in the 24 hours prior to the surgery (Mannitol, Hypertonic saline, Sodium lactate)
* Congestive heart failure
* Moderate ou severe chronic kidney disease, defined by a creatinine clearance (MDRD) < 60 ml/min
* End-stage liver disease (Child Pugh ≥ B7)
* Myasthenia gravis
* External ventricular drain or ventriculoperitoneal shunt of cerebrospinal fluid
* Allergy to Mannitol 20% or one of his excipients
* Allergy to Sodium Lactate or one of his excipients
* Contraindication for propofol
* Allergy to anesthetic agents (propofol, remifentanil, cisatracurium)
* Refusal of consent
* Patient within the exclusion period of another study or planned by the "national file of volunteers"
* Medical history of cognitive disorders or demencia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Quality of brain relaxation | intraoperative
  An adequate brain relaxation is evaluated by the neurosurgeon with a stage 1 (perfectly relaxed) or 2 (acceptably relaxed) of the brain swelling score validated by Todd et al. The brain swelling score is a four-point-scale: 1 (normal brain; no swelling); 2 (minimal swelling, but acceptable); 3 (serious swelling but no specific change in management required); or 4 (severe brain swelling requiring some intervention). Todd et al. reported a significant Relationship between intracranial pressure and the brain swelling score. The brain swelling score is the consensual tool used in clinical trials to assess the clinical effectiveness of brain relaxative therapy.

SECONDARY OUTCOMES:
Necessity for "rescue" therapy | intraoperative
  Proportion of patients who needed a "rescue" therapy in order to improve the brain relaxation and to enable the surgery. "Rescue" therapy consists of the administration of an additional dose of Mannitol 20% 0.25g/kg, deepening the anesthesia (BIS between 20 and 40) or the administration of an intravenous dose of Thiopental 5mg/kg.
Electrolytes alterations | 30 minutes, 60 minutes, 180 minutes, 24 hours and 48 hours after completion of sodium lactate or mannitol infusion
  Variations of natremia (mmol/L), kaliemia (mmol/L), pH and serum osmolarity (mosmol/L) after administration of the osmotherapy.
Changes of lactatemia | 30 minutes, 60 minutes, 180 minutes, 24 hours and 48 hours after completion of sodium lactate or mannitol infusion
  Variations of lactatemia (mmol/L) after administration of the osmotherapy
Volume of post operative brain edema | Day 2 after surgery
  Measurement of the volume of the post operative brain edema by MRI
Glasgow Coma Scale | preoperative, at day 1 and day 2 postoperative
  Assessment of Glasgow coma scale (scale assessing level of conscioussness ranging from 3 = deep unconsciousness to 15 = normal consciousness)
Extubation | Within 2 hours after the end of surgery
  Time between the end of anesthesia and extubation (min)
Neurological recovery | preoperative and Day 2 after surgery
  Neurological revcovery will be assessed comparing the results of a battery of validated neurocognitive tests performed the day before surgery and at Day 2 after surgery.
Protein S100-β | Prior to sodium lactate or mannitol infusion and at 24 hours and at 48 hours after completion of sodium lactate or mannitol infusion
  change in blood level of Protein S100-β
Neuron-Specific Enolase (NSE) | Prior to sodium lactate or mannitol infusion and at 24 hours and at 48 hours after completion of sodium lactate or mannitol infusion
  Change in blood level of Neuron-Specific Enolase (NSE)
Glial Fibrillary Acid Protein (GFAP) | Prior to sodium lactate or mannitol infusion and at 24 hours and at 48 hours after completion of sodium lactate or mannitol infusion
  Change in blood level of Neuron-Specific Enolase (NSE)
Morbidity | Within 30 days after surgery
  Incidence of heart rhythm disorders during the first 48 hours postoperative, intensive care unit length of stay, hospital length of stay, duration of mechanical ventilation, postoperative complications
Mortality | Within 30 days after surgery
  Mortality within 30 days after surgery
Karnofsky performance scale | preoperative and at day 30 after surgery
  The Karnofsky performance scale index is an assessment tool for functional impairment. The lower the Karnofsky score, the worst functional impairment, and in most serious illnesses, the worse likelihood of survival. The Karnofsky performance scale ranges from 0 (dead patient) to 100 (normal no complaints, no evidence of disease).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Todd MM, Warner DS, Sokoll MD, Maktabi MA, Hindman BJ, Scamman FL, Kirschner J. A prospective, comparative trial of three anesthetics for elective supratentorial craniotomy. Propofol/fentanyl, isoflurane/nitrous oxide, and fentanyl/nitrous oxide. Anesthesiology. 1993 Jun;78(6):1005-20. doi: 10.1097/00000542-199306000-00002. PMID 8512094
- [Derived] Besch G, Parmentier AL, Berthier F, Jaeg H, Villeneuve J, Hammoudi F, Scaringella N, Clairet AL, Vettoretti L, Chopard G, Thines L, Ferreira D, Samain E, Pili-Floury S. Clinical effectiveness of hypertonic sodium lactate infusion for intraoperative brain relaxation in patients undergoing scheduled craniotomy for supratentorial brain tumor resection: A study protocol of a single center double-blind randomized controlled phase II pilot trial. Medicine (Baltimore). 2022 Oct 7;101(40):e31038. doi: 10.1097/MD.0000000000031038. PMID 36221362